CLINICAL TRIAL: NCT01131897
Title: Comparative, Randomized, Single-Dose, 2-way Crossover Bioavailability Study of Dr. Reddy's Levetiracetam Tablets, 750 mg and Keppra® 750 mg Tablets of UCB Pharma in Healthy Adult Male Volunteers Under Fasting Conditions.
Brief Title: Bioavailability Study of Levetiracetam Tablets, 750 mg of Dr. Reddy's Under Fasting Conditions.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Mr. M.S. Mohan / Senior Manager - R&D, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AA06179
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Last update posted 2010-06-14 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: Bioavailability; Crossover; Levetiracetam
MeSH Terms: interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levetiracetam (Experimental): Levetiracetam Tablets, 750 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Levetiracetam
- Keppra® (Active Comparator): Keppra® 750 mg Tablets of UCB Pharma Inc.,
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — Levetiracetam Tablets, 750 mg of Dr. Reddy's Laboratories Limited
  Other Names: Keppra® 750 mg Tablets

SUMMARY:
The purpose of this study is to compare the single-dose relative bioavailability study of Levetiracetam Tablets 750 mg with Keppra® 750 mg Tablets under Fasting conditions.

DETAILED DESCRIPTION:
This is an open-label, randomized, single-dose 2-way crossover relative bioavailability study in healthy adult male volunteers under fasting conditions with a washout period of 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male volunteers, 18 to 55 years of age;
* Weighing at least 60 kg and within 15% of their ideal weights (Table of "Desirable Wights of Adults", Metropolitan Life Insurance Company, 1983);
* Medically healthy subjects with clinically normal laboratory profiles and ECGs as deemed by the principal investigator;
* Voluntarily consent to participate in the study

Exclusion Criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease.
* In addition, history or presence of:

  1. alcoholism or drug abuse within the past 2 years;
  2. hypersensitivity or idiosyncratic reaction to levetiracetam;
* Subjects who have been on an special diet (for whatever reason) during the 30 days prior to the first dose and throughout the study.
* Subjects who have made a donation (Standard donation amount or more) of blood or blood products (with the exception of plasma as noted below) within 56 days prior to the first dose.
* Subjects who have made a plasma donation within 7 days prior to the first dose.
* Subjects who have participated in another clinical trial within 30 days prior to the first dose.
* Subjects with hemoglobin less than 12.0 g/dL.
* Subjects who have participated in another clinical trial within 30 days prior to the first dose.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2003-09; Primary Completion 2003-09 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Bioavailability based on Cmax and AUC parameters | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Magdy L Shenouda, MD, Principal Investigator — MDS Pharma Services
Locations (1):
- MDS Pharma Services, Neptune City, New Jersey, United States